CLINICAL TRIAL: NCT06631911
Title: Emotional Awareness and Expression Therapy for Patients With Persistent Physical Symptoms in Routine Psychiatric Care: A Pilot Study
Acronym: EAET for PPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daniel Maroti (Other)
Responsible Party: Sponsor-Investigator, Daniel Maroti, PhD, principal investigator, Stockholm University
Organization: Stockholm University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAET for PPS: a pilot study; 5631 (Other: Signe and Ane Gyllenbergs foundation); 1111 (Other Grant/Funding Number: Prima Psychiatry internal research fund)
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Persistent Physical Symptoms (PPS); Functional Somatic Disorder; Functional Somatic Syndromes; Somatic Symptom Disorder (DSM-5)
Keywords: Emotional Awareness and Expression Therapy; Group psychotherapy; routine care

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotional Awareness and Expression Therapy (Other): Please see description for intervention
  Interventions: Behavioral: Emotional Awareness and Expression Therapy (EAET)

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy (EAET) — Emotional Awareness and Expression Therapy (EAET) is a manualized, short-term psychodynamic therapy that, in this instance, is delivered in a group format.
  The core of Emotional Awareness and Expression Therapy (EAET) involves helping individuals identify, understand, and express their emotions in a therapeutic setting. The therapy emphasizes the connection between unprocessed emotions and physical symptoms, encouraging participants to explore the emotional underpinnings of their distress. Through guided discussions, psychoeducation, and expressive exercises, participants learn to recognize patterns of emotional avoidance, develop self-compassion, and improve interpersonal communication. This process aims to reduce somatic symptoms and enhance overall emotional well-being by fostering a greater awareness of emotional experiences.

SUMMARY:
Emotional Awareness and Expression Therapy (EAET) has emerged as a promising approach for addressing persistent physical symptoms (PPS). Investigating EAET within the context of routine psychiatric care is crucial for several reasons:

Many patients with PPS experience significant distress and functional impairment, yet traditional medical treatments often fail to provide adequate relief. Integrating EAET into routine care could offer a valuable therapeutic option for this population.

Preliminary studies suggest that EAET can lead to significant reductions in pain and other somatic symptoms. Investigating its effectiveness in routine care settings could enhance treatment outcomes for patients who have not responded to conventional therapies.

There is often a disconnect between mental health and physical health treatment in routine care. Investigating EAET can help bridge this gap, fostering collaboration between mental health professionals and primary care providers to address the complexities of patients' health issues.

ELIGIBILITY:
Inclusion Criteria:

* The participant certifies that they have undergone a medical assessment for their physical symptoms (see separate certificate).
* The participant rates either moderate distress from physical symptoms on the PHQ-15 questionnaire (over 10 points) or significant distress from a single physical symptom (at least 2 points for that symptom).
* The participant expresses interest in exploring whether emotional factors, such as stress, may contribute to their symptom profile.
* Any prescribed medications must have been stable for at least one month.

Exclusion Criteria:

* Participants suffer from ongoing substance abuse (alcohol or drugs) or are assessed to have severe mental health issues (psychotic disorders, moderate to high suicide risk, antisocial personality disorder, etc.).
* Participants are currently prescribed medications that are clearly addictive and sedative in nature (e.g., benzodiazepines).
* Participants are involved in other psychological treatments focused on physical symptoms. However, other psychological treatments are permitted as long as the supportive therapy does not occur more than once a month.
* Participants do not have sufficient proficiency in the Swedish language.

Please note that it is the chief physician of each respective research sponsor who, based on collected anamnesis and self-assessment information, makes the final decision regarding whether a participant should be included or excluded from the research project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-15 (PHQ-15) | Pre-post treatment (at treatment termination)
  Somatic symptom severity during the "last week " are assessed with the Patient Health Questionnaire-15 (PHQ-15). Items are rated 0 ("not bothered at all"), 1 ("bothered a little"), or 2 ("bothered a lot"); total scores range from 0 to 30.
Visual Analoge Scales | Pre-post treatment (at treatment termination)
  A second primary outcome is the two Visual Analoge Scales suggested by the EURONET-SOMA network (Rief et al., 2017). Somatic symptom intensity is measured from 1 ("No symptom") to 10 ("Symptom as bad as you can imagine") and somatic symptom interference from 1 ("No interference") to 10 ("Maximum interference").

SECONDARY OUTCOMES:
Sheehan Disability Scale | 1. Pre-post treatment (at treatment termination). 2. Pre-Follow up (12 weeks after intervention).
  SDS consist on three visual analogue scales ranging from 0-10 for symptom interference in daily life. Higher scores indicate worse symptom/functioning, with a maximum score of 30.
Post traumatic symptom Check List-5 (PCL-5), | 1. Pre-post treatment (at treatment termination). 2. Pre-Follow up (12 weeks after intervention).
  PCL-5 consists of 20 questions with ratings 0-4 on impact of post traumatic symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 80.
Patient Health Questionaire-9 (PHQ-9) | 1. Pre-post treatment (at treatment termination). 2. Pre-Follow up (12 weeks after intervention).
  PHQ-9 consists of nine questions withs ratings 0-3 (0= "not at all", 3= "almost every day") on impact of depressive symptoms. Higher scores indicate worse symptom/functioning with a maximum score of 27.
Generalized Anxiety Disorder 7-item scale (GAD-7) | 1. Pre-post treatment (at treatment termination). 2. Pre-Follow up (12 weeks after intervention).
  GAD-7 consists of seven questions with ratings 0-3 (0= "not at all", 3= "almost every day") on impact of anxiety symptoms. Higher scores indicate worse symptom/functioning functioning with a maximum score of 21.
Visual Analoge Scales | Pre-FU (12 weeks after intervention)
  Visual Analoge Scales suggested by the EURONET-SOMA network (Rief et al., 2017). Somatic symptom intensity is measured from 1 ("No symptom") to 10 ("Symptom as bad as you can imagine") and somatic symptom interference from 1 ("No interference") to 10 ("Maximum interference").
Patient Health Questionaire-15 (PHQ-15) | Pre-FU (12 weeks after intervention)
  Somatic symptom severity during the "last week" was assessed with the PHQ-15. Items were rated 0 ("Not bothered at all"), 1 ("Bothered a little"), or 2 ("Bothered a lot"); total scores range from 0 to 30 for women and 0-27 for men.

OTHER OUTCOMES:
Credibility and Expectancy Questionaire (CEQ) | Three weeks into treatment
  The questionnaire consists of several items that participants respond to on a Likert scale (e.g., from 1 to 7), where they rate their level of agreement or belief regarding various statements related to the treatment's credibility and their expected outcomes.
Negative Effects Questionnaire (NEQ) | At FU (12 weeks after intervention).
  The questionnaire includes a series of statements or questions that participants respond to using a Likert scale, where they indicate how often they have experienced these negative effects.
8 visual analgue scales | Mediational measure: Every week during the 12 week long treatment (i.e. 11 measurement points.)
  2 question on 1-10 on symptom intensity and inferference 2 questions on 1-10 on the capacity of self-compassion 2 questions on 1-10 on the capacity of emotional processing 2 question on 1-10 on symptom attribution

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Maroti, PhD, Principal Investigator — Department of Psychology, Faculty of Social Sciences, Stockholm University

IPD SHARING:
Plan to Share IPD: No
The participants has not agreed to this